CLINICAL TRIAL: NCT03834727
Title: Characterizing the Impact and Treatment of Reproductive Tract Bleeding on Women and Post-menarchal Girls With Bleeding Disorders.
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: American Thrombosis and Hemostasis Network (Network)
Responsible Party: Principal Investigator, Kristina Haley, Associate Professor, Oregon Health and Science University
Other Study IDs: 00018857
Record Dates: First submitted 2018-12-18; First posted 2019-02-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Hemophilia A; Bleeding Disorder
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Characterizing the impact and treatment of reproductive tract bleeding on women and post-menarchal girls with bleeding disorders.

Objectives: This is a cross-sectional observational study of women and girls (WG) with bleeding disorders enrolled in the American Thrombosis and Hemostasis Network (ATHN) dataset. Based on the investigators' study of currently available data of WG with bleeding disorders in the ATHNdataset, the investigators hypothesize that the information currently captured in the core data elements of the ATHNdatasest does not adequately capture data specific to WG with bleeding disorders. Further, the investigators hypothesize that it is feasible for Hemophilia Treatment Centers (HTCs) to include data points specific to WG with bleeding disorder when enrolling participants in the ATHNdataset. This hypothesis will be evaluated through the following specific aims:

Specific Aim 1: Characterize reproductive tract bleeding in a cohort of WG with bleeding disorders cared for at US HTCs.

Specific Aim 2: Characterize the treatment strategies for and the impact of heavy menstrual bleeding in a cohort of females with bleeding disorders cared for at HTCs.

Specific Aim 3: Evaluate the feasibility of adding female specific core data points to the ATHNdataset.

DETAILED DESCRIPTION:
This is a multi-center, cross-sectional study of women and girls with bleeding disorders receiving care at Hemophilia Treatment Centers (HTCs). To further characterize this population, WG who receive care at federally funded US HTCs will be approached regarding participation. Following assent and/or consent, participants will be asked to complete a series of forms. In order to assess their bleeding symptoms, they will complete the self-BAT (Bleeding Assessment Tool) as well as the Menstrual Bleeding Questionnaire (MBQ). In order to assess their quality of life, they will complete the PROMIS-29 quality of life inventories. Patients may be contacted if they miss a question on any of these forms. Phone call should take no more than 15 minutes. Study staff will complete an intake form which includes data regarding bleeding disorder diagnosis as well as treatment, using information obtained from the patient, chart review, and the ATHNdataset.

ELIGIBILITY:
Inclusion Criteria:

* Women and girls with an active diagnosis of a congenital bleeding disorder (as designated by the institution inputting data);

  1. Deficiencies of factors VIII, IX, II, V, VII, VII, IX, X, XI, FV+VIII, XIII, Plasminogen Activator Inhibitor 1(PAI-1), hypo-, a-, or dys-fibrinogenemia
  2. von Willebrand Disease (Type 1, Type 1c, Type 2A, Type 2B, Type 2M, Type 2N, Type 3, Low VWF)
  3. Any platelet function disorder (i.e. Glanzmann Thrombasthenia, Bernard Soulier Syndrome, Platelet Storage Pool disorder, MYH9 disorders, Gray Platelet syndrome, Dense granule deficiency)
  4. Ehlers Danlos Syndrome
* Post-menarchal: has had at least 1 period at the time of study entry
* Participating in the ATHNdataset

Exclusion Criteria:

* Male gender
* Acquired bleeding disorder
* Thrombotic disorder
* Non-English speaking

Ages: 10 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women and girls receiving care at federally funded US Hemophilia Treatment Centers will be approached regarding participation.
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Reproductive tract bleeding will be characterized utilizing the ISTH-BAT(International Society of Thrombosis and Haemostasis Bleeding Assessment Tool) | 1 year
  The ISTH-BAT is the International Society on Thrombosis and Hemostasis Bleeding Assessment Tool and can be self-administered. It provides an overall bleeding score as well as information about specific bleeding symptoms.
Reproductive tract bleeding will be characterized utilizing the Menstrual Bleeding Questionnaire. | 1 year
  The Menstrual Bleeding Questionnaire is a patient reported outcome tool specific to the symptom of menstrual bleeding. It is also self-administered.
Reproductive tract bleeding will be characterized by reviewing the medical history | 1 year
  Utilizing the current ATHNdataset data forms, the medical history will be reviewed and symptoms and diagnoses specific to menstrual bleeding will be entered.
Identify treatment strategies for heavy menstrual bleeding through patient report | 1 year
  Utilizing a form previously developed, participants will indicate previous treatments utilized for heavy menstrual bleeding and rank their effectiveness.
Evaluate impact through quality of life tool (PROMIS-29) | 1 year
  Participants will complete the PROMIS-29 quality of life tool.
Evaluate impact through quality of life tool (EQ-5D) | 1 year
  Participants will complete the EQ-5D quality of life tool.
Evaluate the feasibility of entering female specific core data points to the ATHNdataset. | 1 year
  Study site coordinators will complete a feasibility questionnaire regarding the challenges of adding female specific data to the ATHNdataset.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Haley, DO, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States